CLINICAL TRIAL: NCT03468179
Title: Acute Effects of Dietary Oatmeal on Serum Levels of N-acyl-phosphatidylethanolamines and Their Metabolites.
Brief Title: Oatmeal Effect on N-acyl-phosphatidylethanolamines
Acronym: NAPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Sean Davies, Associate Professor, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: JJWPending
Record Dates: First submitted 2018-03-09; First posted 2018-03-16 (Actual); Results first posted 2019-12-13 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-11

CONDITIONS: Obesity; Cardiovascular Diseases
Keywords: Diet; N-acyl-phosphatidylethanolamine; N-acyl-ethanolamine; NAPE; NAE; Oatmeal
MeSH Terms: conditions — Obesity; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: All subjects will have baseline blood drawn, fed controlled serving of oatmeal, and blood drawn sequentially over subsequent 2 hours.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Oatmeal (Experimental): Subjects will arrive for study fasting. IV access will be obtained, and baseline blood drawn. They will be fed 80gm/100kg oatmeal, and blood levels will be drawn at 30, 60, 90, and 120 minutes.
  Interventions: Dietary Supplement: Oatmeal

INTERVENTIONS:
Dietary Supplement: Oatmeal — Subjects will be fed a calculated serving of oatmeal.

SUMMARY:
N-acyl-phosphatidylethanolamine (NAPEs) and their active metabolites, N-acyl-ethanolamides (NAEs) are lipid satiety factors that are normally biosynthesized in the intestinal tract in response to food intake. Reduced levels of NAPEs and NAEs have been found in obese individuals, and increasing plasma NAPE and NAEs levels may be beneficial to obese individuals trying to lose weight or to keep off weight gain after losing weight. We have found that oatmeal has large amounts of NAPEs, and based on previous mouse studies, we hypothesize that a single dose of dietary oatmeal is sufficient to double plasma NAE from baseline, possibly inducing satiety and increasing basal metabolic rate. To test this hypothesis, we will feed volunteers a single weight-based serving of oatmeal while monitoring its effects on serum glucose, NAPE and NAE levels as well as on subjective satiety.

DETAILED DESCRIPTION:
N-acyl-phosphatidylethanolamine (NAPEs) and their active metabolites, N-acyl-ethanolamides (NAEs) are lipid satiety factors that are normally biosynthesized in the intestinal tract in response to food intake. Reduced levels of NAPEs and NAEs have been found in obese individuals, so that increasing plasma NAPE and NAEs levels may be beneficial to obese individuals trying to lose weight or to keep off weight gain after losing weight. While NAPEs are endogenously synthesized by mammals in their intestinal tract, many other organisms, including plants, also biosynthesize NAPEs. Recent screening of a wide range of foods by our lab demonstrated that oatmeal (Regular Instant Oatmeal) had very large amounts of NAPEs (0.17 mg NAPE / g dry oatmeal), suggesting that consumption of oatmeal may be a straightforward mechanism for elevating plasma NAPE and NAE levels in obese individuals. Based on our previous mouse studies with synthetic NAPE and with bacteria biosynthesizing NAPE, we hypothesize that a dose of oatmeal sufficient to deliver 0.135 mg NAPE per kg body should be sufficient to double plasma NAE levels from baseline, thereby inducing satiety and increasing basal metabolic rate. For a 100 kg person, 80 grams of dry regular instant oatmeal (2 servings) provides this 0.135 mg / kg dose. (The dose of dry oatmeal per person = (body weight in kg / 100 kg)* 80 g dry oatmeal. Thus for 50 kg person, 40 g dry oatmeal (1 serving) provides the required dose.) This amount of dry oatmeal is converted to the test meal by adding sufficient water to overtop oatmeal by about 1 cm (or to consistency desired by volunteer) and then microwaving for ~3-4 minutes on high. In the initial testing, no additives such as butter, cream, or brown sugar should be used in preparation or serving oatmeal. Water can be consumed ad lib.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* non-pregnant
* normal BMI (20-25)

Exclusion Criteria:

* Obese
* underweight
* diabetes mellitus
* coronary artery disease
* oatmeal allergies
* hyper/hypocoagulability
* food intolerances
* Irritable bowel syndrome
* Inflammatory bowel disease
* Celiac disease
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — 5 Male, 5 female
Enrollment: 10 (Actual)
Dates: Start 2018-10-07 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sean Davies, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oatmeal
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Oatmeal: Participants will be fed 80gm/100kg oatmeal, and blood levels will be drawn at 30, 60, 90, and 120 minutes.
  Oatmeal: Subjects will be fed a calculated serving of oatmeal.
Arm/Group | Oatmeal
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum N-acyl-phosphatidylethanolamine (NAPE)
Description: Change in serum NAPE from baseline to 120 minutes post-oatmeal challenge
Time Frame: Baseline to 120 minutes
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Oatmeal
Number analyzed (Participants) | 10
nmol/L | -4.02 (10.57)

2. Secondary Outcome: Serum NAPE
Description: Serum NAPE Levels at 30, 60, and 90 minutes
Time Frame: 30, 60, and 90 minutes
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Oatmeal
Number analyzed (Participants) | 10
nmol/L
  30 minutes | 3.36 (7.38)
  60 minutes | 2.78 (4.17)
  90 minutes | 4.12 (7.71)

3. Secondary Outcome: Serum N-acyl-ethanolamides (NAE)
Description: Serum NAE levels at baseline, 30, 60, 90 and 120 minutes
Time Frame: baseline 30, 60, 90 and 120 minutes
Population: 5 participants had pre and post NAE levels below the level of detection for reasons that were unclear
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Oatmeal
Number analyzed (Participants) | 5
nmol/L
  Baseline | 0.09 (0.02)
  30 minutes | 0.08 (0.012)
  60 minutes | 0.07 (0.013)
  90 minutes | 0.06 (0.010)
  120 minutes | 0.07 (0.009)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for each participant for 1 study day.
Description: Adverse events used clinical.trials.gov definitions.
Arm/Group | Oatmeal
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oatmeal (N=10)
light-headed / dizziness (Injury, poisoning and procedural complications) | 1 (1) — patient became lightheaded during IV placement, resolved with rest, able to complete study.

LIMITATIONS AND CAVEATS:
Limitation of this study was that only 1 dose of oatmeal was used and the study group was relatively small.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2018-07-02): https://cdn.clinicaltrials.gov/large-docs/79/NCT03468179/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2018-07-06): https://cdn.clinicaltrials.gov/large-docs/79/NCT03468179/Prot_SAP_001.pdf